CLINICAL TRIAL: NCT07093099
Title: Efficacy of Enhanced Focused Education and Counseling on Adequacy of Mechanical Bowel Preparation Among High-Risk Patients: A Randomized Clinical Trial
Brief Title: Effect of Counseling and Education on Mechanical Bowel Preparation
Acronym: EEFEC-AMBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Ram Drug Store (Industry)
Collaborators: An-Najah National University (Other)
Responsible Party: Principal Investigator, Mohammed M. H. Hajhamad, MB, BCH (Egypt) DoS (Malaysia) Consultant Surgeon and Endoscopist Head of Department of Continuous Medical Education and Clinical Research - Rafidia Surgical Hospital, An-Najah National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/134/162; 2021/134/162 (Other: Palestinian MOH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Colonoscopy; Colorectal Cancer Screening
Keywords: Bowel prep; Colonoscopy preparation; BBPS (Boston Bowel Preparation Scale); Enhanced education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Endoscopists scoring bowel preparation using the Boston Bowel Preparation Scale (BBPS) were blinded to the participant's group assignment. Participants and care providers were not masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Education Group (Experimental): Participants in this group received enhanced bowel preparation education. The intervention included:
  Face-to-face counseling by trained staff about the importance of bowel prep and how to follow instructions; A 6-minute instructional video explaining dietary restrictions, purgative usage, and procedure timeline; A printed booklet with illustrated step-by-step instructions; and Access to a smartphone app with automated reminders, preparation tracking, and guidance.
  All participants used the same bowel cleansing agent (polyethylene glycol-based preparation).
  Interventions: Behavioral: Enhanced Education Package for Bowel Preparation; Other: Standard Education Leaflet
- Standard Education Group (Active Comparator): Participants in this group received standard bowel preparation instructions in the form of a hospital-issued informational leaflet. This leaflet included basic written instructions about dietary restrictions, timing and method of laxative use, and preparation day logistics.
  No counseling, video, or app-based support was provided. The same bowel cleansing agent was used in both arms.
  Interventions: Other: Standard Education Leaflet

INTERVENTIONS:
Behavioral: Enhanced Education Package for Bowel Preparation — a multifaceted intervention was designed to improve mechanical bowel preparation (MBP) in patients undergoing colonoscopy. It included:
  Structured face-to-face counseling on the importance of bowel prep, potential complications of poor prep, and how to follow instructions.
  A 6-minute instructional video explaining step-by-step dietary and medication instructions.
  A printed booklet with visual aids summarizing key steps.
  A mobile phone app delivering interactive reminders, tracking tools, and preparation guidance.
  All participants used the same polyethylene glycol-based bowel cleansing agent.
  Other Names: Enhanced Counseling; Video Instruction; Booklet and Mobile App Support
  Arms: Enhanced Education Group
Other: Standard Education Leaflet — Participants in this arm received a standard hospital-issued bowel preparation instruction leaflet. The document provided written instructions on dietary modifications, timing and dosage of the bowel cleansing agent, and day-of-procedure guidance. No personalized counseling, video support, or reminder tools were provided. This reflects the routine care practice at the study hospitals.
  Other Names: Standard Instructions; Usual Care Preparation

SUMMARY:
The goal of this clinical trial is to learn whether enhanced education and counseling can improve bowel preparation before colonoscopy in high-risk patients. The main questions it aims to answer are:

Does enhanced education lead to better bowel cleansing as measured by the Boston Bowel Preparation Scale (BBPS)?

Does it improve patient satisfaction, compliance with instructions, and procedure efficiency?

Researchers will compare an enhanced education program (including counseling, video, booklet, and mobile app) to standard written instructions typically given before colonoscopy.

Participants will:

Be randomly assigned to either the enhanced education group or the standard instruction group

Undergo routine colonoscopy after following the assigned preparation method

Complete short questionnaires about their experience, satisfaction, and willingness to repeat the process

This study is being done at two hospitals in Palestine.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Undergoing elective colonoscopy

Considered high-risk for inadequate bowel preparation, including at least one of the following:

Prior abdominal or pelvic surgery

Chronic constipation (fewer than 3 bowel movements per week)

Use of constipating medications (e.g., opioids, tricyclic antidepressants, calcium channel blockers)

Age >65 years

Multiple comorbidities (e.g., diabetes, neurologic disorders affecting motility)

----------------------------------------------------

Exclusion Criteria:

Known allergy or intolerance to bowel preparation agents

Pregnancy

Severe comorbidities (e.g., decompensated liver disease, severe heart failure)

Cognitive impairment or illiteracy preventing understanding of instructions

Emergency colonoscopy or known obstructive colorectal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) Total Score | During the procedure itself
  The BBPS is a validated scoring system to assess bowel cleanliness during colonoscopy. It ranges from 0-9, with three sub-scores (right, transverse, left colon) each scored 0-3. Higher scores indicate better bowel preparation quality. Total BBPS score will be compared between groups.

SECONDARY OUTCOMES:
Patient Satisfaction Score | Within 24 hours after colonoscopy
  Measured on a 10-point Likert scale, with 1 = very dissatisfied and 10 = very satisfied. Participants were surveyed about their experience with the preparation process.
Cecal Intubation Time | During the procedure itself
  Time (in minutes) from insertion of the colonoscope to successful intubation of the cecum, recorded by the performing endoscopist. Lower times indicate more efficient procedures.
Willingness to Repeat Preparation | Within 24 hours after colonoscopy
  Participant-reported willingness to use the same bowel preparation method again, expressed as a binary outcome (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed M Hajhamad, MD, Principal Investigator — An-Najah National University
Locations (1):
- Rafidia Surgical Hospital, Nablus, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No